CLINICAL TRIAL: NCT03075280
Title: Pre-ERCP Carbohydrate Drinks Improve Patients Recovery: an ERAS Protocol Attempts in ERCP
Brief Title: Pre-ERCP High Carbohydrate Drinks Improve Patients Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Xun Li, M.D., Ph. D, Direct of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSIGansu
Record Dates: First submitted 2017-03-04; First posted 2017-03-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Complication
Keywords: ERCP; ERAS; complication; fatigue; high carbohydrate diet
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High carbohydrate liquid diet (Experimental): No need preoperative fasting more than 6 hours. Uptake 400ml high carbohydrate liquid diet 2 hours before ERCP.
  Interventions: Procedure: 400ml high carbohydrate liquid diet before ERCP
- Routine ERCP group (No Intervention): Preoperative fasting more than 6 hours as usual.

INTERVENTIONS:
Procedure: 400ml high carbohydrate liquid diet before ERCP — 400ml high carbohydrate liquid diet uptake 2 hours before ERCP
  Other Names: Routine ERCP
  Arms: High carbohydrate liquid diet

SUMMARY:
To test the benefits of extra high carbohydrate liquid diet uptake 2 hours before ERCP in improving patients' early recovery.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) has been formed of procedure which contains preoperative education, improvement of anesthesia, reducing the number of drainage tubes, and early diet after surgery. In recent years, because of its positive advantages, ERAS was widely accepted in surgical fields.

For upper gastrointestinal surgery, high-carbohydrate drinks can be given 2 hours before surgery in order to guarantee the stability of blood glucose and circulation during the operation. It obviously reduce the preoperative thirst, hunger, irritability and even the incidence of postoperative complications.

However ERAS program is rarely studied in ERCP. Theoretically we can use ERAS as a strategy to reduce post-ERCP uncomfortable and complications.

ELIGIBILITY:
Inclusion Criteria:

* ERCP patients,
* Age 18-85 years old.

Exclusion Criteria:

* Coagulation dysfunction (INR> 1.3) and low peripheral blood platelet count(<50×109 / L) or using anti-coagulation drugs,
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage, severe liver disease, shock, liver or kidney malfunction,
* Diabetes（blood glucose fluctuations）or with complications,
* Intestinal obstruction or other contraindications with feeding and watering,
* Prior surgery of Bismuth Ⅱ and Roux-en-Y,
* Pregnant women,
* Unwillingness or inability to consent for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1292 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
Levels of fatigue (Fatigue Scale-14 scoring system) | 6 months
  The patients always feel tired and faint. The clinical manifestation includes slow to respond, the flexibility and coordination disorders.
Abdominal pain | 6 months
  Pain score (scores:1-10)

SECONDARY OUTCOMES:
The average incubation time | 6 months
  The time of total procedure
Successful cannulation time | 6 months
  From first achieve the papilla to success cannulation
Postoperative abdominal distention | 6 months
  Distention uncomfortable
Postoperative nausea and vomiting | 6 months
  Nausea or vomiting after procedure
Complications | 6 months
  Pancreatitis, cholangitis, bleeding, aspiration, et,al.
Blood glucose | 6 months
  Intra-operative blood glucose and 2 hours' blood glucose after procedure
Intraoperative residues in stomach | 6 months
  The volume of stomach residues
The time eating | 6 months
  The time of eager to eat after procedure
Length of hospital stay | 6 months
  Days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, M.D., Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (15):
- China (15):
  - Third Military Medical University, Chongqing, Chongqing Municipality
  - The first hospital of Lanzhou university, Lanzhou, Gansu
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tongji medical collage,Huazhong University of science and technology, Wuhan, Hubei
  - Second Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yingchuan, Ningxia
  - The first affiliated hospital of Xi 'an jiaotong university, Xi'an, Shaanxi
  - Shandong jiaotong Hospital, Jinan, Shandong
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Taiyuan Iron and Steel Corporation Hospital, Taiyuan, Shanxi
  - Tianjin Nankai Hospital, Tianjin, Tianjin Municipality
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Shulan Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meng W, Leung JW, Wang Z, Li Q, Zhang L, Zhang K, Wang X, Wang M, Wang Q, Shao Y, Zhang J, Yue P, Zhang L, Zhu K, Zhu X, Zhang H, Hou S, Cai K, Sun H, Xue P, Liu W, Wang H, Zhang L, Ding S, Yang Z, Zhang M, Weng H, Wu Q, Chen B, Jiang T, Wang Y, Zhang L, Wu K, Yang X, Wen Z, Liu C, Miao L, Wang Z, Li J, Yan X, Wang F, Zhang L, Bai M, Mi N, Zhang X, Zhou W, Yuan J, Suzuki A, Tanaka K, Liu J, Nur U, Weiderpass E, Li X. Safety of high-carbohydrate fluid diet 2 h versus overnight fasting before non-emergency endoscopic retrograde cholangiopancreatography: A single-blind, multicenter, randomized controlled trial. Chin Med J (Engl). 2024 Jun 20;137(12):1437-1446. doi: 10.1097/CM9.0000000000002820. Epub 2023 Aug 24. PMID 37620294